CLINICAL TRIAL: NCT05728138
Title: Culturally Adapted Psychosocial Intervention for Suicidal Ideation in Individuals With First Episode Psychosis: A Feasibility Randomised Controlled Trial
Brief Title: Psychosocial Intervention for Suicidal Ideation in Individuals With FEP: A Feasibility Trial
Acronym: CMAP-FEP
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Pakistan Institute of Living and Learning (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SAHAR M-CMAPPlus FEP 07
Record Dates: First submitted 2023-02-04; First posted 2023-02-14 (Actual); Last update posted 2025-01-03 (Actual); Status verified 2025-01

CONDITIONS: Self Harm, First Episode Psychosis
Keywords: Self-harm, First Episode Psychosis, adaptation, problem-solving.
MeSH Terms: conditions — Self-Injurious Behavior

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CMAP Plus FEP (Experimental): Participants with First episode of psychosis, Culturally Adapted Manual Assisted Problem Solving (CMAP) integrated with Culturally adapted Cognitive Behavior Therapy (CaCBT)
  Interventions: Behavioral: CMAP Plus CBT
- treatment as usual (No Intervention): Participants in this group will continue their routine treatment as prescribed by their responsible clinician. In Pakistan TAU mostly comprise of antipsychotics with few patients having access to psychological therapies. Research staff will record the nature and intensity of the TAU for each participant

INTERVENTIONS:
Behavioral: CMAP Plus CBT — Culturally Adapted Manual Assisted Problem Solving (CMAP) integrated with Culturally adapted Cognitive Behavior Therapy (CaCBT) CMAP is a manual assisted brief psychological intervention based on the principles of Cognitive Behaviour Therapy (CBT), integrated with Culturally adapted Cognitive Behavior Therapy (CaCBT) including 12 sessions delivered over three months. This intervention includes evaluation of the self-harm attempt, psycho-education, crisis skills, problem-solving and simple and thought management
  Arms: CMAP Plus FEP

SUMMARY:
To check the feasibility and acceptability of Culturally adapted Cognitive Behavioral Therapy for Psychosis (CaCBTp) and Culturally Adapted Manual Assisted Brief Psychological Intervention for Self-harm (CMAP), which we have provisionally called (CMAP Plus) for individuals experiencing Suicidal Ideation (SI) in First Episode Psychosis (FEP).

DETAILED DESCRIPTION:
Psychosis is one of the 20 leading causes of disability worldwide, affecting 29 million people. First Episode Psychosis (FEP) occurs at a young age and is thought to be a critical period, influencing the long-term course of the disorder. The early course of psychosis is characterised by repeated relapses with up to 80 % relapsing within five years of an initial episode. It has been reported that individuals diagnosed with psychosis disorders are also identified with developing experiences of self-harm, completed suicide or suicide attempt. A systematic review on identification of correlation between self-harm/suicidality and FEP, also suggested association of suicidal ideation or self-injurious behavior though additional research is highly recommended in this particular subject Psychological therapies are widely used in the high-income countries, but very limited in LMIC like Pakistan due to factors including lack of trained mental health workers and inadequate infrastructure to support secondary mental health services. These factors, amongst others, contribute to the significant treatment gap in LMICs like Pakistan. There are currently no early intervention services in Pakistan and given the shortage of appropriately trained clinicians to deliver psychosocial interventions novel approaches are needed. We have culturally adapted Cognitive Behavior therapy which demonstrated feasibility and acceptability for psychosis in Pakistan. To address suicide specific symptoms, content will be integrated from the life after self-harm manual (CMAP. It is a CBT based problem solving intervention for self-harm which has been adapted in Pakistan in a feasibility trial and a recently completed MRC funded large multicenter trial (n=901)

ELIGIBILITY:
Inclusion Criteria:

* Individuals diagnosed with, Schizophrenia or Schizoaffective disorder according to DSM-V, confirmed by treating consultant.
* Age 18 and above years able to understand written and spoken Urdu.
* A score of 1 (Mild- Frequent thoughts of being better off dead, or occasional thoughts of suicide.) on the Calgary depression Scale item 8 (Suicide) "Have you felt that life wasn't worth living? Did you ever feel like ending it all? What did you think you might do? Did you actually try?"
* Individuals with a score of 3 or more on any of the positive symptoms on the Positive and Negative Syndrome Scale (PANSS) (e.g., delusions, hallucination).

Exclusion Criteria:

* Any evidence of organic brain disease, clinically significant comorbid illness or learning disability. Participants deemed actively suicidal by their designated health professional.
* Those scoring >1 on Calgary depression Scale will be excluded and be referred to a psychiatric service.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2023-11-01 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-10-30 (Estimated)

PRIMARY OUTCOMES:
Feasibility Indicator | From baseline to 12th week (end of intervention)
  feasibility will be determined by collecting data on recruitment and retention rates.
  The success criterion of feasibility will be to recruit > 50% of eligible participants
Acceptability Indicator | From baseline to 12th week (end of intervention)
  Intervention acceptability will be assessed using data on attendance. Criterion for acceptability is a mean attendance rate of >70%.

SECONDARY OUTCOMES:
Positive and Negative Syndrome Scale | From baseline to 12th week (end of intervention)
  The Scale will examine the Positive and Negative Syndrome for Schizophrenia and is comprised of 30 items. The 30 items of semi structured questionnaire will measure positive syndromes, like delusions, hallucinations, and conceptual disorganisation whereas negative syndromes include passive or apathetic social avoidance and blunted affect. It will also indicate the magnitude of relation to one another and to psychopathology in generic term (e.g., anxiety, guilt, depression, and lack of insight).
Beck Scale for Suicidal Ideation | From baseline to 12th week (end of intervention)
  This is a 19-item instrument for detecting and measuring the thoughts of an individual that they might want to kill him/herself during the past week. This scale has been used with schizophrenia, schizoaffective, or bipolar disorders
Medication Adherence Rating Scale | From baseline to 12th week (end of intervention)
  We will use MARS to check adherence to medications. MARS is a 10-item measure. It incorporates features of both the Drug Attitude Inventory (DAI) and the Morisky Medication Adherence Scale (MMAS). The patient will be asked to choose the answer which best describes their behaviour or attitude towards their medication during the past week.
Calgary Depression Scale | From baseline to 12th week (end of intervention)
  The scale is specially designed to measure the depression for Psychosis, consist of nine items. CDS will indicate the subjective and qualitative dimensions of depression in Schizophrenia
The Work and Social Adjustment Scale | From baseline to 12th week (end of intervention)
  Five items scale that measures the perceived impairment of social life, relationships, home management, work and private leisure having scores between 0 to 8 that means 0 (no impairment) and 8 (very severe impairment) with a total score of 40
EuroQol-5 Dimensions EQ5-D | From baseline to 12th week (end of intervention)
  Quality of life will be measured in five dimensions, including usual activities, anxiety/depression, pain/discomfort, self-care, and mobility.
Client Service Receipt Inventory | From baseline to 12th week (end of intervention)
  The information will be collected on the use of other health services such as (faith healers/Imams) using CSRI.

CONTACTS AND LOCATIONS:
Overall Officials: Imran Chaudhry, Principal Investigator — Ziauddin Hospital
Locations (1):
- Karwan e Hayat, Karachi, Sindh, Pakistan

IPD SHARING:
Plan to Share IPD: No